CLINICAL TRIAL: NCT05130866
Title: A Two-staged, Phase 2/3, Randomized, Multicenter Study to Evaluate the Efficacy and Safety of REC-2282 in Participants With Progressive NF2 Mutated Meningiomas
Brief Title: Efficacy and Safety of REC-2282 in Patients With Progressive Neurofibromatosis Type 2 (NF2) Mutated Meningiomas
Acronym: POPLAR-NF2
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to sponsor decision. This decision was not related to safety concerns with REC-2282.
Sponsor: Recursion Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-2282-201
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Neurofibromatosis Type 2
Keywords: Neurofibromatosis Type 2; Neurofibromatosis Type II
MeSH Terms: conditions — Neurofibromatosis 2 | interventions — HDAC-42

STUDY DESIGN:
Intervention Model Description: A Two-staged, Phase 2/3, Randomized, Multicenter Efficacy and Safety Study.
Who Masked: Participant, Investigator
Masking Description: Masking applies to Cohort B only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A Adults, REC-2282 40 mg (Experimental): Adult participants will receive REC-2282.
  Interventions: Drug: REC-2282
- Cohort A Adults, REC-2282 60 mg (Experimental): Adult participants will receive REC-2282.
  Interventions: Drug: REC-2282
- Cohort A Adolescents, REC-2282 (Experimental): Adolescent participants will receive REC-2282.
  Interventions: Drug: REC-2282
- Cohort B REC-2282 (Experimental): Participants will receive REC-2282.
  Interventions: Drug: REC-2282
- Cohort B Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REC-2282 — Participants will receive REC-2282 3 times per week orally for 3 weeks followed by 1 week off for a 4-week cycle.
  Other Names: AR-42; OSU-HDAC42; NSC-D736012
  Arms: Cohort A Adolescents, REC-2282; Cohort A Adults, REC-2282 40 mg; Cohort A Adults, REC-2282 60 mg; Cohort B REC-2282
Drug: Placebo — Participants will receive placebo orally 3 times per week for 3 weeks followed by 1 week off for a 4-week cycle.
  Arms: Cohort B Placebo

SUMMARY:
This is a two-staged, Phase 2/3, randomized, multi-center study to investigate the efficacy and safety of REC-2282 in participants with progressive NF2 mutated meningiomas.

DETAILED DESCRIPTION:
Cohort A (Phase 2) will provide early data on efficacy and safety of REC-2282 in participants with progressive NF2 mutated meningiomas, and provide guidance for the dose in the confirmatory part of the study (Cohort B, Phase 3). The purpose of Cohort B of the study is to assess the efficacy and safety of REC-2282 compared with placebo in participants with progressive NF2 mutated meningiomas.

In both cohorts, there will be a screening period of up to 8 weeks, a treatment period, a 4-week safety follow-up period after the end of treatment, and a 6-month post-study follow-up. The first 8 participants enrolled in Cohort A will complete a food effect run-in sub study. At the end of the study period, participants may be offered participation in an open-label extension (OLE) period.

In Cohort A, adult participants will be randomized to one of two dose levels of REC-2282.

In Cohort B, participants will be randomized to REC-2282 treatment (dose to be determined from Cohort A) arm or placebo arm in a ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

1. ≥12 years of age and weighing at least 40 kg
2. Progressive meningioma that is amenable to volumetric analysis
3. Has either 1) sporadic meningioma with confirmed NF2 mutation; or, 2) confirmed diagnosis of NF2 disease (revised Manchester criteria); or, 3) at least one NF2-related tumor (with pathogenic germline or proven mosaic NF2 variant)
4. Adequate bone marrow function
5. Has provided written informed consent/assent to participate in the study

Exclusion Criteria:

1. Progressive disease associated with significant or disabling clinical symptoms likely to require surgery or radiation therapy within the next 3 months.
2. Received prior surgery, radiosurgery, or laser interstitial thermal therapy in the target tumor, or immediately adjacent to the target tumor within 12 months prior to screening.
3. Received an anti- tumor agent for meningioma within 3 months, or 5 half-lives (whichever is longer), prior to screening.
4. History of an active malignancy within the previous 3 years except for localized cancers that are considered cured, and, in the opinion of the investigator, present a low risk of recurrence.
5. Received another investigational drug within 30 days prior to screening
6. Pregnant, lactating, or is planning to attempt to become pregnant or impregnate someone during this study or within 90 days after the last dosing cycle.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Cohort A: Number of Participants with Progression-free survival (PFS) at 6 Months | 6 months
  In Cohort A, PFS is defined as the number of participants who are alive and progression-free at 6 months with progression defined as having an increase of 20% or more in the target tumor identified.
Cohort B: Number of Participants with PFS up to 3 years | Up to 3 years
  In Cohort B, PFS is defined as the time from the date of randomization until disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Cohort A: Change from Baseline in Target Tumor Volume at 6 Months | 6 months
Cohort A: Number of Participants with PFS at 12 and 24 Months | 12 and 24 Months
  In Cohort A, PFS is defined as the number of participants who are alive and progression-free at 12 and 24 months with progression defined as having an increase of 20% or more in the target tumor identified.
Cohorts A and B: Objective Response Rate (ORR) | Up to 3 years
Cohorts A and B: Disease Control Rate (DCR) | Up to 3 years
Cohorts A and B: Time to Response (TTR) | Up to 3 years
Cohorts A and B: Duration of Response (DOR) | Up to 3 years
Cohorts A and B: Time to Surgery/radiation for Target Tumors | Up to 3 years
Cohorts A and B: Maximum Observed Plasma Concentration (Cmax) of REC-2282 | Up to 3 years
Cohorts A and B: Time to Maximum Plasma Concentration (Tmax) of REC-2282 | Up to 3 years
Cohorts A and B: Area under the curve from 0 to 24hr (AUC) of REC-2282 | Predose to 24 hours postdose

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - House Institute, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Sarah Cannon Cancer Institute - HCA Midwest, Overland Park, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota / Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No